CLINICAL TRIAL: NCT03265223
Title: Randomized Controlled Study of Intraincisional Infiltration Versus Intraperitoneal Instillation of Standardized Dose of Ropivacaine 0.2% in Post-laparoscopic Cholecystectomy Pain
Brief Title: Ropivacaine Use Intraincisionally Versus Intraperitoneally for Post-Laparoscopic Cholecystectomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jawaharlal Nehru Medical College (Other)
Responsible Party: Principal Investigator, Kaushal Deep Singh, Principal Investigator, Jawaharlal Nehru Medical College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JawaharlalNMC
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Ropivacaine; Laparoscopic Cholecystectomy; Pain
Keywords: Ropivacaine; local anesthesia; intraincisional infiltration; intraperitoneal instillation; post-laparoscopic cholecystectomy pain; shoulder pain; rescue analgesia; triple blinding
MeSH Terms: conditions — Pain; Shoulder Pain | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Three study groups: Controls received no drug, intraperitoneal group received drug along right hemidiaphragm and in gallbladder fossa while intraincisional group received drug by infiltration at trocar site
Who Masked: Participant, Care Provider, Investigator
Masking Description: Triple blinding was done i.e. neither the operating surgeon nor the investigator and nor the patient knew to which study group patient belong to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Controls (No Intervention): Received 1 ml/cm normal saline (23 ml) both at intraperitoneal (=20 ml) as well as intraincisional (=3 ml) location.
- Intraperitoneal group (Active Comparator): Received 20 ml of 0.2% ropivacaine intraperitoneally (1 ml/cm; 16 ml along right hemi-dome, approximately equal to length of right hemi-dome of diaphragm in an average adult and 4 ml in gall bladder fossa) and 3 ml normal saline (1ml/cm of port site incision length)
  Interventions: Drug: 0.2% ropivacaine
- Intraincisional group (Active Comparator): Received 20 ml of normal saline intraperitoneally (1 ml/cm; 16 ml along right hemi-dome, approximately equal to length of right hemi-dome of diaphragm in an average adult and 4 ml in gall bladder fossa) and 3 ml 0.2% ropivacaine (1ml/cm of port site incision length)
  Interventions: Drug: 0.2% ropivacaine

INTERVENTIONS:
Drug: 0.2% ropivacaine — Intraperitoneal instillation versus intraincisional infiltration
  Other Names: Ropin; Naropin
  Arms: Intraincisional group; Intraperitoneal group

SUMMARY:
Pain still remains a limiting factor in early discharge of patients undergoing laparoscopic cholecystectomy. Almost all earlier studies done to compare the efficacy of local anaesthetics used intraperitoneally as compared to intraincisionally used equal amounts of drugs at the two locations, usually 10-20 ml. Using this large amount of drug in the small space of intraincisional location as compared to similar amount of drug in large intraperitoneal space created an inadvertent bias in favor of patients receiving the drug intraincisionally so such patients naturally experienced less pain. The investigators decided to standardize the drug used at these two locations as 1ml/cm and conduct a new study comparing the effects of drugs in relieving pain when used at these two locations.

DETAILED DESCRIPTION:
Aims & Objectives: To conduct a randomized, triple-blind, placebo-controlled study by standardizing dose of local anesthetic, to compare the effectiveness of intraperitoneal against intraincisional use of ropivacaine 0.2% for post-laparoscopic cholecystectomy pain relief.

Materials & Methods: American Society of Anesthesiologists (ASA) physical status I or II patients underwent elective 4 port laparoscopic cholecystectomy by a single surgeon. Anesthetic and surgical techniques were standardized. Patients were randomized using envelope method into 3 groups according to location of drug use. Triple blinding was ensured and envelopes were opened only at the completion of study. All patients received ~23 ml of solution, of which 20 ml was given intraperitoneally [1 ml/cm; 16 ml along right hemi-dome, approximately equal to length of right hemi-dome of diaphragm in an average adult and 4 ml in gall bladder fossa) and ~3 ml intraincisionally (1 ml/cm of length of incision). Controls (n=86) received ~23 ml normal saline (20 ml intraperitoneally and 1 ml/cm intraincisionally) while the intraperitoneal group (n=100) received 20 ml of intraperitoneal instillation of injection ropivacaine 0.2% and 1 ml/cm of normal saline intraincisionally at the end of procedure. Intraincisional group (n=108) received 20 ml normal saline intraperitoneally and 1 ml/cm of injection ropivacaine 0.2% infiltration at incisional site at the end of procedure. All patients received injection diclofenac sodium 75mg/1ml (aqueous) intravenously 12 hourly postoperatively. 5 different pain scales were used for assessment of overall pain. Pain scores were assessed at 5 points of time, that is, at 0.5, 4, 8, 12 and 24 hours postoperatively. Shoulder pain and extra dose of analgesic required (rescue analgesia) were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients in the age group of 15-80 years
* Patients conferring to Grade I or II of American Society of Anesthesiologists (ASA) physical status classification system only
* Patients undergoing elective Laparoscopic Cholecystectomy
* Patients having symptomatic cholelithiasis only
* Patients operated by a single surgeon were included.

Exclusion Criteria:

* Patients with known allergic reactions to local anesthetics
* Cases that were converted to open cholecystectomy
* Patients with major intra-operative complications
* Patients suffering from acute cholecystitis, empyema or malignancy of gall bladder, having history of chronic pain or those taking frequent analgesics or opioids pre-operatively
* Patients with peptic ulceration, bleeding disorders, impaired renal and/or hepatic function, and sensitivity to NSAIDs or opioids.
* Patients in whom gall bladder (GB) stones are found incidentally on ultrasonography (USG) (asymptomatic cholelithiasis)
* Patients suffering from severe chronic medical diseases and morbid obesity
* Patients unable to comprehend instructions or having communication problems were excluded from the study.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 353 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Effect of ropivacaine use intraincisionally versus intraperitoneally as compared to controls on post-laparoscopic cholecystectomy pain | 36 months
  To study and assess the effect and impact of using the local anesthetic ropivacaine 0.2%, over controls, on the intensity of postoperative pain in patients undergoing laparoscopic cholecystectomy; and to compare and assess the optimal site i.e. intraincisional versus intraperitoneal of using local anesthetic (ropivacaine) for better post-laparoscopic cholecystectomy pain relief.

SECONDARY OUTCOMES:
Identify the component of pain which is dominant after undergoing laparoscopic cholecystectomy | 36 months
  To identify the component of pain (visceral versus incisional component) that is dominant after laparoscopic cholecystectomy; and after how much interval of time it assumes importance?
Laparoscopic cholecystectomy as day-case using ropivacaine only | 36 months
  To strive for making laparoscopic cholecystectomy a truly day case procedure in the public setup of developing countries like India by using this cheap local anaesthetic alone
Changing trends in epidemiology of cholelithiasis | 36 months
  To check for any changing trends in epidemiology of cholelithiasis in North India

CONTACTS AND LOCATIONS:
Overall Officials: Kaushal D Singh, MS Surgery, Principal Investigator — Jawaharlal Nehru Medical College, Aligarh

IPD SHARING:
Plan to Share IPD: Undecided
Data of those patients will be shared patients who will give consent for the same.

DOCUMENTS (3):
  • Study Protocol (2014-04-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT03265223/Prot_000.pdf
  • Informed Consent Form (2014-04-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT03265223/ICF_001.pdf
  • Statistical Analysis Plan (2014-04-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT03265223/SAP_002.pdf